CLINICAL TRIAL: NCT04332133
Title: Anatomical and Functional Outcomes of Subthreshold Micropulse Laser Versus Intravitreal Ranibizumab Injection in Treatment of Diabetic Macular Edema
Brief Title: Outcomes of Subthreshold Laser Versus Intravitreal Injection of Ranibizumab in Diabetic Macular Edema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Raafat Mohyeldeen Abdelrahman Abdallah, associate professor of ophthalmology, Minia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Diabetic Macular Edema(DME)
Record Dates: First submitted 2020-03-30; First posted 2020-04-02 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Diabetic Macular Edema
Keywords: DME, mfERG, SML, ranibizumab,IV.injection
MeSH Terms: interventions — Intravitreal Injections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group 1 (Active Comparator): group 1 of DME which treated by SML
  Interventions: Procedure: laser interference,INTRAVITREAL INJECTION
- group 2 (Active Comparator): Group 2 of DME which treated by intravitreal injection of Ranibizumab
  Interventions: Procedure: laser interference,INTRAVITREAL INJECTION
- group 3 (No Intervention): control group of diabetic patients received no treatment

INTERVENTIONS:
Procedure: laser interference,INTRAVITREAL INJECTION — sub threshold micro pulse laser for DME for group 1 and intravitreal injection of Ranibizumab for group 2
  Arms: group 1; group 2

SUMMARY:
The aim of this study is To compare the anatomical and functional results of intravitreal( IV) injection of ranibizumab with sub threshold micropulse laser ( SML) in treatment of Diabetic macular edema (DME) both anatomically by spectral domain optical coherence tomography (SD OCT) and functionally by best-corrected visual acuity (BCVA) and multifocal electroretinogram (mfERG).

DETAILED DESCRIPTION:
Diabetic macular edema (DME) causes significant visual loss in diabetic patients. About 20% and 40% of patients with Type 1 and Type 2 diabetes mellitus (DM), respectively, develop DME. One-third of diabetic patients who have had DM for more than twenty years will develop DME . Early impairment in the function of the middle and inner layers of the retina has been reported in diabetic patients before appearance of vascular complications . A good independent guide of macular function in patients with DME is multifocal electroretinogram (mfERG) readings from the macular area, which strongly associate with morphologic alterations in the macula. Some investigators suggested that temporal characteristic (implicit time) of mfERG waves are more important than amplitudes for evaluation of retinal function in diabetic patients. They concluded that patients with DM show temporal changes indicating delayed neural transmission due to local impairment of blood glucose metabolism. In contrast, others emphasize the importance of both parameters (implicit time and amplitude) in identifying retinal affection in DM.

Intravitreal (IV) injections of anti-vascular endothelial growth factor (VEGF) agents provided good visual outcomes in treatment of DME. However, IV anti-VEGF injections are expensive, need to be repeated many times and have the potential risk of causing endophthalmitis . Subthreshold micropulse laser (SML) treatment of DME has the same effect as conventional laser treatment, nonetheless, there is less damage to adjacent tissues of the burn area in the retinal pigment epithelium (RPE). SML allows laser emission to be divided into bursts of short cyclic pulses that remain for microseconds permitting substantial cooling amid these short pulses .

ELIGIBILITY:
Inclusion Criteria:

* DME with BCVA<0.5 decimal Snellen acuity.
* Controlled blood glucose (HbA1c) <6.5%.

Exclusion Criteria:

* History of previous intraocular surgery,
* History of previous laser treatment,
* History of previous IV injection,
* Macular disease or ischemia,
* Proliferative diabetic retinopathy,
* Vitreoretinal traction,
* Interruption of external limiting membrane (ELM) or ellipsoid zone (EZ).
* Dense media opacity,
* Optic disc pathology
* History of strokes or ischaemic heart diseases.
* patients with (CST) > 400 µm on OCT .

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
central subfield thickness in micrometer | 6 months
  OCT for the macular area with measuring CST in micron
p1 amplitude of mfERG | 6mnths
  p1 amplitude of multifocal ERG measured in nv/deg2
BCVA | 6 months
  BCVA is measured in decimal of Snellen visual acuity

CONTACTS AND LOCATIONS:
Overall Officials: Raafat Abdallah, A.professor, Principal Investigator — ophthalmology department,faculty of medicine, minia university; Mahmoud Genidy, professor, Study Director — ophthalmology department,faculty of medicine, minia university; Wagiha Massoud, professor, Study Chair — ophthalmology department,faculty of medicine, minia university

IPD SHARING:
Plan to Share IPD: Yes
The results can be shred after the end of the work.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: after publication has been completed
Access Criteria: personal communication through email or through this site if possible

REFERENCES:
- [Background] Klein R, Knudtson MD, Lee KE, Gangnon R, Klein BE. The Wisconsin Epidemiologic Study of Diabetic Retinopathy XXIII: the twenty-five-year incidence of macular edema in persons with type 1 diabetes. Ophthalmology. 2009 Mar;116(3):497-503. doi: 10.1016/j.ophtha.2008.10.016. Epub 2009 Jan 22. PMID 19167079
- [Background] Lung JC, Swann PG, Wong DS, Chan HH. Global flash multifocal electroretinogram: early detection of local functional changes and its correlations with optical coherence tomography and visual field tests in diabetic eyes. Doc Ophthalmol. 2012 Oct;125(2):123-35. doi: 10.1007/s10633-012-9343-0. Epub 2012 Jul 25. PMID 22828871
- [Background] Yamamoto S, Yamamoto T, Hayashi M, Takeuchi S. Morphological and functional analyses of diabetic macular edema by optical coherence tomography and multifocal electroretinograms. Graefes Arch Clin Exp Ophthalmol. 2001 Feb;239(2):96-101. doi: 10.1007/s004170000238. PMID 11372551
- [Background] Fortune B, Schneck ME, Adams AJ. Multifocal electroretinogram delays reveal local retinal dysfunction in early diabetic retinopathy. Invest Ophthalmol Vis Sci. 1999 Oct;40(11):2638-51. PMID 10509661
- [Derived] Abdelrahman A, Massoud W, Elshafei AMK, Genidy M, Abdallah RMA. Anatomical and functional outcomes of subthreshold micropulse laser versus intravitreal ranibizumab injection in treatment of diabetic macular edema. Int J Retina Vitreous. 2020 Dec 3;6(1):63. doi: 10.1186/s40942-020-00265-6. PMID 33292788